CLINICAL TRIAL: NCT06103292
Title: Ionized Calcium Level Abnormalities In Major Trauma Patients Pre And Post Receiving Blood Transfusion And Its Relation To Mortality Rate
Brief Title: Calcium Levels in Major Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hossam Abdel Rahman Ahmed Ismail (Other)
Responsible Party: Sponsor-Investigator, Hossam Abdel Rahman Ahmed Ismail, Hossam Ismail, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Calcium abnormaities in trauma
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Major Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ionized calcium levels — measuring calcium level in trauma patients

SUMMARY:
To assess and treat The calcium level abnormalities in major trauma pre and post receiving blood transfusions .

DETAILED DESCRIPTION:
Primary objective:

* to evaluate the level of ionized calcium in multiple trauma patients with massive hemorrhage

Secondary objective:

* to build a relation between the level of ionized calcium and the degree of hemorrhagic shock

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old - < 70 years
2. Major trauma patients.
3. Admission and Ionized calcium measurement before blood transfusions

Exclusion Criteria:

1. patients below 18 years or > 70 years of age.
2. Pregnant women
3. Arrested patients
4. Patients managed outside the hospital and had received blood transfusions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study all consecutive adult multiple trauma patients presenting to the emergency department with the inclusion criteria until the sample size is satisfied.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
follow up ionized calcium level | 24 hrs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauaia A, Moore FA, Moore EE, Moser KS, Brennan R, Read RA, Pons PT. Epidemiology of trauma deaths: a reassessment. J Trauma. 1995 Feb;38(2):185-93. doi: 10.1097/00005373-199502000-00006. PMID 7869433
- [Background] Heckbert SR, Vedder NB, Hoffman W, Winn RK, Hudson LD, Jurkovich GJ, Copass MK, Harlan JM, Rice CL, Maier RV. Outcome after hemorrhagic shock in trauma patients. J Trauma. 1998 Sep;45(3):545-9. doi: 10.1097/00005373-199809000-00022. PMID 9751548
- [Background] Zink KA, Sambasivan CN, Holcomb JB, Chisholm G, Schreiber MA. A high ratio of plasma and platelets to packed red blood cells in the first 6 hours of massive transfusion improves outcomes in a large multicenter study. Am J Surg. 2009 May;197(5):565-70; discussion 570. doi: 10.1016/j.amjsurg.2008.12.014. PMID 19393349
- [Background] Barry GD. Plasma calcium concentration changes in hemorrhagic shock. Am J Physiol. 1971 Apr;220(4):874-9. doi: 10.1152/ajplegacy.1971.220.4.874. No abstract available. PMID 5551141